CLINICAL TRIAL: NCT07144527
Title: Nicotinamide Mononucleotide Supplementation for Exercise Tolerance Improvement in Healthy Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Scott Silveira (Other)
Collaborators: Concordia University Chicago (Other); EGACeutical (Unknown)
Responsible Party: Sponsor-Investigator, Scott Silveira, Principle Investigator, Concordia University Chicago
Organization: Concordia University Chicago (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2305604-1
Record Dates: First submitted 2025-08-19; First posted 2025-08-27 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Aging; Frailty; Exercise Tolerance; Healthy Male and Female Subjects
Keywords: Nicotinamide Mononucleotide; NAD+ Metabolism; Exercise Tolerance; Aging; Older Adults; Betaine; Hydrogen Peroxide (low-dose, dietary); High Intensity Interval Training; VO2peak; Lactate Threshold; Critical Power; Anaerobic Work Capacity; Healthy Volunteers
MeSH Terms: conditions — Frailty | interventions — Betaine; Hydrogen Peroxide; Nicotinamide Mononucleotide

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind trial with two parallel groups, each using a two-period crossover design. One group receives EGA and a placebo in a random sequence, and the other group receives NMN and a placebo in a random sequence.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1 - EGA -> Placebo (Experimental): Participants receive EGA during Period 1, followed by Placebo during Period 2 after a washout. Assigned Interventions: EGA; Placebo.
  Interventions: Dietary Supplement: NMN, betaine, low-dose hydrogen peroxide (EGA); Dietary Supplement: Placebo
- Arm 2 - Placebo -> EGA (Experimental): Participants receive Placebo during Period 1, followed by EGA during Period 2 after a washout. Assigned Interventions: Placebo; EGA.
  Interventions: Dietary Supplement: NMN, betaine, low-dose hydrogen peroxide (EGA); Dietary Supplement: Placebo
- Arm 3 - NMN -> Placebo (Experimental): Participants receive Nicotinamide Mononucleotide (NMN) during Period 1, followed by Placebo during Period 2 after a washout. Assigned Interventions: NMN; Placebo.
  Interventions: Dietary Supplement: Nicotinamide Mononucleotide (NMN); Dietary Supplement: Placebo
- Arm 4 - Placebo -> NMN (Experimental): Participants receive Placebo during Period 1, followed by NMN during Period 2 after a washout. Assigned Interventions: Placebo; NMN.
  Interventions: Dietary Supplement: Nicotinamide Mononucleotide (NMN); Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: NMN, betaine, low-dose hydrogen peroxide (EGA) — Proprietary formulation containing NMN, betaine, and low-dose hydrogen peroxide.
  Arms: Arm 1 - EGA -> Placebo; Arm 2 - Placebo -> EGA
Dietary Supplement: Nicotinamide Mononucleotide (NMN) — Conventional NMN supplement.
  Arms: Arm 3 - NMN -> Placebo; Arm 4 - Placebo -> NMN
Dietary Supplement: Placebo — Organoleptically matched inert control.

SUMMARY:
This is a randomized, double-blind, placebo-controlled, two-arm crossover clinical trial evaluating the effects of a patented age-reversal therapy, EGA®, compared to conventional nicotinamide mononucleotide (NMN) supplementation. The study will assess safety and efficacy in improving exercise tolerance and modulating biomarkers of aging in healthy older adults.

The primary outcome is cycle ergometry constant work rate (CWR) exercise tolerance, measured as time to fatigue. Secondary outcomes include changes in peak oxygen consumption (VO₂peak), critical power, anaerobic work capacity, lactate threshold, and NAD⁺ metabolite levels.

EGA® is composed of three metabolomic compounds that are endogenous to humans. The formulation has been used in prior exploratory studies and real-world applications, which have helped inform the design of this current trial.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled, two-arm crossover trial will compare the effects of two NAD⁺-modulating interventions-EGA® and conventional nicotinamide mononucleotide (NMN) supplementation-on exercise tolerance and metabolic biomarkers in healthy older adults. EGA® is a proprietary formulation composed of three endogenously occurring metabolomic compounds (including NMN) and has been used in prior non-FDA-regulated studies involving human participants. The EGA® arm will involve a twice-daily oral dose of EGA® containing 1000 mg of NMN, while the comparison arm will involve twice-daily oral dose of 1000 mg of conventional NMN per day. Doses will be self-administered each morning and evening with water.

The primary endpoint is time to fatigue during constant work rate cycle ergometry (CWR-Tlim), a validated surrogate for submaximal exercise tolerance. Secondary endpoints include peak oxygen uptake (VO₂peak), lactate threshold, anaerobic work capacity, and critical power, in addition to circulating NAD⁺ and its related metabolites.

The trial is designed to evaluate the short-term physiological effects and biological activity of EGA® compared to conventional NMN under tightly controlled exercise testing and training conditions. Data from this study will be used to inform the therapeutic potential of EGA® in improving physical performance in healthy older adults (60-80 years). Future directions may include further clinical evaluation or regulatory submissions, depending on outcomes from this pilot investigation.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 60 to 80 years, of any sex
* Written clearance from primary care physician confirming medical fitness to participate in an exercise-based clinical study
* Normal or near-normal cardiovascular function to safely engage in moderate to vigorous exercise, demonstrated by either: stress echocardiogram or coronary CT angiogram within the past 12 months showing normal left ventricular function, no significant valvular heart disease, no ischemic changes, and no other clinically significant abnormalities, plus confirmation that no new cardiovascular symptoms (e.g., chest pain, dyspnea, syncope) or changes in health status have occurred since testing
* Montreal Cognitive Assessment (MoCA) score of 26 or higher
* Free from acute or uncontrolled chronic medical conditions that would pose a risk or interfere with study participation
* Physically capable of engaging in structured exercise involving moderate to vigorous intensity stationary cycling
* Successful completion of a graded exercise test (e.g., stationary bike) without significant adverse events or contraindications
* Ability to attend at least four in-person laboratory visits in Beverly Hills, California
* Non-smoker for at least 12 months
* Able to provide informed consent and comply with study procedures
* Willing to refrain from initiating new exercise, dietary supplement, or medication regimens during the study

Exclusion Criteria:

* Severe cardiovascular disease (e.g., recent myocardial infarction <6 months, unstable angina, uncontrolled hypertension >160/100 mmHg)
* Severe respiratory conditions (e.g., advanced COPD or other conditions preventing exercise participation)
* Significant neurological impairments that hinder comprehension of instructions or participation in exercise
* Terminal illness or conditions limiting life expectancy or ability to complete the study
* Severe cognitive impairment preventing informed consent, protocol adherence, or comprehension of interventions
* Significant orthopedic limitations or injuries that prevent safe exercise participation
* Use of NMN, NR, or other NAD+-altering supplements within the past 14 weeks
* Anticipated or current alcohol consumption >2 drinks per week, or unwillingness to abstain from alcohol during the study
* Current substance abuse affecting study participation or adherence
* Other acute or chronic health conditions judged by the investigators to pose risk or interfere with study objectives
* Non-compliance with study requirements, withdrawal of informed consent, or unforeseen circumstances compromising completion
* Any condition which, in the opinion of the investigator, would interfere with study participation or interpretation of results

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Time to Fatigue During Constant Work Rate Cycle Ergometry (tLIM). | Measured at the beginning and end of each 4-week intervention period.
  Duration (in seconds) that participants can sustain a constant submaximal workload on a cycle ergometer until volitional fatigue. This is a validated surrogate for submaximal exercise tolerance.

SECONDARY OUTCOMES:
Peak Oxygen Uptake (VO2max) | Measured at the beginning and end of each 4-week intervention period.
  Maximum oxygen consumption (ml/kg/min) achieved during graded exercise testing.
Lactate Threshold | Measured at the beginning and end of each 4-week intervention period.
  Workload or oxygen consumption corresponding to the point at which blood lactate concentration rises above baseline, assessed via graded exercise testing and gas exchange sampling.
Anaerobic Work Capacity | Measured at the beginning and end of each 4-week intervention period.
  Cumulative work performed above the critical power, calculated from cycle ergometer testing.
Critical Power | Measured at the beginning and end of each 4-week intervention period.
  The asymptote of the power-duration relationship. A work rate reflecting sustainable aerobic work capacity.
Circulating NAD+ and Related Metabolites | Measured at the beginning and end of each 4-week intervention period.
  Plasma concentrations of NAD+, NMN, and related metabolites measured by targeted metabolomics.

OTHER OUTCOMES:
Adverse Events | From first dose through final study visit (up to 12 weeks per participant, including two 4-week intervention periods and a 4-week washout).
  Incidence of any reported adverse events or side effects during intervention periods.
Adherence to Supplementation | Assessed weekly during each 4-week intervention period and at the end of each intervention period (Weeks 4 and 12), for a total study duration of up to 12 weeks per participant.
  Pill counts and participant self-report logs of study product usage.
Exercise Session Adherence | Assessed weekly during each 4-week intervention period and summarized at the end of each period (Weeks 4 and 12); total study duration up to 12 weeks per participant.
  Proportion of prescribed exercise sessions completed (percentage of sessions completed (%) per intervention period, verified by attendance log.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Office of Dr. Robert Huizenga MD, Beverly Hills, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the primary and secondary outcome results reported in this study will be shared. This includes data related to exercise testing outcomes (tLIM, VO2max, lactate threshold, anaerobic work capacity, critical power) and metabolomics (circulating NAD+ and related metabolites). Demographic and baseline characteristics will also be included in de-identified form.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD and supporting information will be available within 12 months of publication of the primary results and will remain available for 5 years thereafter.
Access Criteria: Data will be made available to qualified researchers upon submission of a methodologically sound research proposal. Requests should be directed to the Principal Investigator, and access will be granted after review and approval by the study steering committee. Data will be shared under a data use agreement to ensure participant confidentiality.